CLINICAL TRIAL: NCT05935254
Title: Comparative Evaluation of Plaque Removal Efficacy of Electric Toothbrushes Between Children With Attention Deficit And Hyperactivity Disorder And Healthy Children
Brief Title: Plaque Removal Efficacy of Electric Toothbrushes in ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Melis AKYILDIZ, Assistant Professor Bahar Melis AKYILDIZ, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AdnanMU-ZUCAR.001
Record Dates: First submitted 2023-03-06; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Attention Deficit and Hyperactivity Disorder; Dental Plaque
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADHD-Electric Toothbrush Group (Experimental): Children aged 8-10 years who were diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) according to DSM-5 criteria, who applied to Aydın Adnan Menderes University Faculty of Medicine Child Psychiatry Clinic, were randomly assigned to the electric toothbrush group.
  Interventions: Device: Plaque removal efficacy of children's electric toothbrush (Oral-B D100 Vitality; Procter & Gamble, Cincinnati, OH, United States)
- ADHD-Manual Toothbrush Group (Experimental): Children aged 8-10 years who were diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) according to DSM-5 criteria, who applied to Aydın Adnan Menderes University Faculty of Medicine Child Psychiatry Clinic, were randomly assigned to the manual toothbrush group.
  Interventions: Device: Plaque removal efficacy of children's soft manual toothbrush (Oral-B Stages 6-12 years; Procter & Gamble, Cincinnati, OH, United States)
- Healthy- Electric Toothbrush Group (Active Comparator): Among the physically and psychologically healthy children aged 8-10 who applied to the Pediatric Dentistry Clinic of ADU Faculty of Dentistry, those assigned to the electric toothbrush group as a result of randomization
  Interventions: Device: Plaque removal efficacy of children's electric toothbrush (Oral-B D100 Vitality; Procter & Gamble, Cincinnati, OH, United States)
- Healthy- Manual Toothbrush Group (Active Comparator): Among the physically and psychologically healthy children aged 8-10 who applied to the Pediatric Dentistry Clinic of ADU Faculty of Dentistry, those assigned to the manual toothbrush group as a result of randomization
  Interventions: Device: Plaque removal efficacy of children's soft manual toothbrush (Oral-B Stages 6-12 years; Procter & Gamble, Cincinnati, OH, United States)

INTERVENTIONS:
Device: Plaque removal efficacy of children's electric toothbrush (Oral-B D100 Vitality; Procter & Gamble, Cincinnati, OH, United States) — At the baseline appointment, Löe-Silness Gingival Index values were recorded in all fully erupted permanent teeth and primary teeth without exfoliation. Mira-2-Ton Plaque Staining Solution was applied to the labial and lingual surfaces of all teeth with a micro brush to determine the amount of dental plaque before the first brushing. After plaque discoloration, the Approximal Plaque Index and the Turesky Modification of Quigley-Hein Plaque Index values were recorded. The children brushed their teeth with an electric toothbrush for 2 minutes, under the supervision of a physician who was not included in the study. Plaque discoloration was performed again to determine the amount of plaque removal after the first brushing. Approximal Plaque Index and The Turesky modification of the Quigley-Hein Plaque Index the measurements were recorded. The same procedures were repeated to evaluate the brushing habits at the 1st-month and 3rd-month, respectively.
  Arms: ADHD-Electric Toothbrush Group; Healthy- Electric Toothbrush Group
Device: Plaque removal efficacy of children's soft manual toothbrush (Oral-B Stages 6-12 years; Procter & Gamble, Cincinnati, OH, United States) — At the baseline appointment, Löe-Silness Gingival Index values were recorded in all fully erupted permanent teeth and primary teeth without exfoliation. Mira-2-Ton Plaque Staining Solution was applied to the labial and lingual surfaces of all teeth with a micro brush to determine the amount of dental plaque before the first brushing. After plaque discoloration, the Approximal Plaque Index and the Turesky Modification of Quigley-Hein Plaque Index values were recorded. The children brushed their teeth with a manual toothbrush for 2 minutes, under the supervision of a physician who was not included in the study. Plaque discoloration was performed again to determine the amount of plaque removal after the first brushing. Approximal Plaque Index and The Turesky modification of the Quigley-Hein Plaque Index the measurements were recorded. The same procedures were repeated to evaluate the brushing habits at the 1st-month and 3rd-month, respectively.
  Arms: ADHD-Manual Toothbrush Group; Healthy- Manual Toothbrush Group

SUMMARY:
A total of 52 children, 26 of whom were diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) as the experimental group and 26 healthy with no systemic disease as the control group, were included in the study. Then, in order to evaluate the effectiveness of electric and manual toothbrushes, each group was randomly divided into 2 subgroups: Electric and Manual. Children were educated on toothbrushing according to subgroups. DMFT/dft and Löe-Silness Gingival Index (GI) values were recorded. At the first appointment, plaque disclosing was performed and Turesky modification of Quigley-Hein Plaque Index (TQHPI) and Approximal Plaque Index (API) values were recorded to determine the amount of dental plaque before the brushing. Subsequently, children brushed their teeth for 2 minutes with the subgroup's toothbrush type. Then, plaque disclosing and measurements were repeated to determine the amount of plaque removal after brushing. The same procedure steps were repeated at the 1st and 3rd-month appointments, respectively. a p-value below 0.05 was considered statistically significant.

DETAILED DESCRIPTION:
A total of 52 children, 26 of whom were diagnosed with ADHD, as the experimental group and 26 of whom were healthy, as the control group, were included in the study. Intraoral examination of the children was performed in a dental chair. Standard coding systems and tools developed by the World Health Organization were used to collect data in calculating the criteria for oral health. Soft tissues, tongue, cheek, and palate area were checked in each examination period. Intraoral examination was performed carefully, from the distal right maxillary molars to the most distal right mandibular molars. If there was no cavitation with white spot lesions and black/dark and bright discolorations were considered healthy. According to the DMFT index (Decayed, Missing, and Filled Teeth Index) with the obtained records, DMFT values for permanent teeth and dft values for primary teeth were calculated.

Randomization of the patients to determine the subgroups was carried out by the physician who performed the first examination (B.M.A) using a computer program called www.Random.org (Randomness and Integrity Services Ltd., Ireland). In order to evaluate the effectiveness of electric and manual toothbrushes, each group was divided into 2 subgroups according to the types of brush (electric and manual). There are a total of 4 subgroups in the study. In the manual toothbrush subgroups, the children had a demonstration of how to brush with the Bass Technique on the model. The electric toothbrush subgroups had a demonstration about how to brush their teeth with an electric toothbrush according to the manufacturer's instructions on the model. During the study, children brushed their teeth at home under parental supervision. It is instructed to brush teeth for 2 minutes 2 times a day. During the study period, Sensodyne Promine Kids (GlaxoSmithKline Brazil Ltda, Jacarepagua, Rio de Janeiro, Brazil) were given to children. In both the experimental and control groups and their parents had received instruction to avoid oral hygiene procedures such as flossing and using mouthwash during the study period, except tooth brushing.

After randomization, at the first appointment, Löe-Silness Gingival Index values were recorded in all fully erupted permanent teeth and primary teeth without exfoliation. In order to determine the amount of dental plaque before the first brushing, Mira-2-Ton Plaque Staining Solution (Hager Werken, Germany) was applied to the labial and lingual surfaces of all teeth with a micro brush, and then the children were asked to rinse their mouths with water for 30 seconds. After plaque discoloration, the Approximal Plaque Index and the Turesky Modification of Quigley-Hein Plaque Index values were recorded. The children brushed their teeth in front of a mirror for 2 minutes with the toothbrushes according to subgroups, under the supervision of a physician who was not included in the study. To determine the amount of plaque removal after the first brushing, plaque discoloration was performed again. The Turesky modification of the Quigley-Hein Plaque Index and the Approximal Plaque Index measurements were recorded. The same procedures were repeated to evaluate the brushing habits at the 1st-month and 3rd-month, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Having not had oral prophylaxis in the last 1 month
* Taking not antibiotics within the last 1 month
* Having not had severe periodontal disease and dental caries
* Having no pain symptoms due to caries in any of their teeth,
* Not using any orthodontic appliances
* Not using an electric toothbrush before
* Having at least 16 teeth in the mouth

Exclusion Criteria:

* Have a complex medical history
* Have psychiatric illness other than attention deficit and hyperactivity disorder

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Determination of Gingival Index (GI) values | The measurements will be done before the intervention at baseline
  Evaluation of children's gingival health during the study period
Determination of Gingival Index (GI) values | The measurements will be done before the intervention at 1st month
  Evaluation of children's gingival health during the study period
Determination of Gingival Index (GI) values | The measurements will be done before the intervention at 3rd month
  Evaluation of children's gingival health during the study period
Determination of Turesky modification of Quigley-Hein Plaque Index (TQHPI) values | The measurements will be done immediately before the intervention at baseline
  Evaluation of plaque removal efficiency from labial and lingual surfaces of teeth with a toothbrush
Determination of Turesky modification of Quigley-Hein Plaque Index (TQHPI) values | The measurements will be done immediately after the intervention at baseline
  Evaluation of plaque removal efficiency from labial and lingual surfaces of teeth with a toothbrush
Determination of Turesky modification of Quigley-Hein Plaque Index (TQHPI) values | The measurements will be done immediately before the intervention at 1st month
  Evaluation of plaque removal efficiency from labial and lingual surfaces of teeth with a toothbrush
Determination of Turesky modification of Quigley-Hein Plaque Index (TQHPI) values | The measurements will be done immediately after the intervention at 1st month
  Evaluation of plaque removal efficiency from labial and lingual surfaces of teeth with a toothbrush
Determination of Turesky modification of Quigley-Hein Plaque Index (TQHPI) values | The measurements will be done immediately before the intervention at 3rd month
  Evaluation of plaque removal efficiency from labial and lingual surfaces of teeth with a toothbrush
Determination of Turesky modification of Quigley-Hein Plaque Index (TQHPI) values | The measurements will be done immediately after the intervention at 3rd month
  Evaluation of plaque removal efficiency from labial and lingual surfaces of teeth with a toothbrush
Determination of Approximal Plaque Index (API) values | The measurements will be done immediately before the intervention at baseline
  Evaluation of plaque removal efficiency from proximal surfaces of teeth with a toothbrush
Determination of Approximal Plaque Index (API) values | The measurements will be done immediately after the intervention at baseline
  Evaluation of plaque removal efficiency from proximal surfaces of teeth with a toothbrush
Determination of Approximal Plaque Index (API) values | The measurements will be done immediately before the intervention at 1st month
  Evaluation of plaque removal efficiency from proximal surfaces of teeth with a toothbrush
Determination of Approximal Plaque Index (API) values | The measurements will be done immediately after the intervention at 1st month
  Evaluation of plaque removal efficiency from proximal surfaces of teeth with a toothbrush
Determination of Approximal Plaque Index (API) values | The measurements will be done immediately before the intervention at 3rd month
  Evaluation of plaque removal efficiency from proximal surfaces of teeth with a toothbrush
Determination of Approximal Plaque Index (API) values | The measurements will be done immediately after the intervention at 3rd month
  Evaluation of plaque removal efficiency from proximal surfaces of teeth with a toothbrush

SECONDARY OUTCOMES:
Determination of the DMFT Index (Decayed, Missing and filled Teeth Index) of the subgroups | Baseline
  To determine the risk of dental caries in the permanent dentition period of children during the study period.
Determination of the DMFT Index (Decayed, Missing and filled Teeth Index) of the subgroups | 3rd Month
  To determine the risk of dental caries in the permanent dentition period of children during the study period.
Determination of the dft Index (decay filled teeth index) of the subgroups | Baseline
  To determine the risk of dental caries in the primary dentition of children during the study period.
Determination of the dft Index (decay filled teeth index) of the subgroups | 3rd Month
  To determine the risk of dental caries in the primary dentition of children during the study period.
A questionnaire consisting of 19 questions that all children participating in the study could answer with their parents. | Baseline
  To determine of nutrition, diet, and tooth brushing habits of children and sociodemographic factors

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Melis AKYILDIZ, Study Director — Aydın Adnan Menderes University, Turkey; Zeynep UÇAR, Principal Investigator — Aydın Adnan Menderes University, Turkey; Aylin Kaya, Principal Investigator — Aydın Adnan Menderes University, Turkey
Locations (1):
- Aydın Adnan Menderes University Faculty of Dentistry Department of Pediatric Dentistry, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polanczyk GV, Salum GA, Sugaya LS, Caye A, Rohde LA. Annual research review: A meta-analysis of the worldwide prevalence of mental disorders in children and adolescents. J Child Psychol Psychiatry. 2015 Mar;56(3):345-65. doi: 10.1111/jcpp.12381. Epub 2015 Feb 3. PMID 25649325
- [Background] Drumond VZ, Souza GLN, Pereira MJC, Mesquita RA, Amin M, Abreu LG. Dental Caries in Children with Attention Deficit/Hyperactivity Disorder: A Meta-Analysis. Caries Res. 2022;56(1):3-14. doi: 10.1159/000521142. Epub 2021 Dec 20. PMID 34929707
- [Background] Paszynska E, Krahel A, Pawinska M, Dmitrzak-Weglarz M, Perczak A, Slopien A, Gawriolek M. Management for Caries Prevention in ADHD Children. Int J Environ Res Public Health. 2022 Jun 17;19(12):7455. doi: 10.3390/ijerph19127455. PMID 35742701
- [Background] Atmetlla G, Burgos V, Carrillo A, Chaskel R. Behavior and orofacial characteristics of children with attention-deficit hyperactivity disorder during a dental visit. J Clin Pediatr Dent. 2006 Spring;30(3):183-90. doi: 10.17796/jcpd.30.3.g66h2750h11242p6. PMID 16683663
- [Background] Pirila-Parkkinen K, Pirttiniemi P, Nieminen P, Tolonen U, Pelttari U, Lopponen H. Dental arch morphology in children with sleep-disordered breathing. Eur J Orthod. 2009 Apr;31(2):160-7. doi: 10.1093/ejo/cjn061. Epub 2008 Nov 20. PMID 19028674
- [Background] Andersson H, Sonnesen L. Sleepiness, occlusion, dental arch and palatal dimensions in children attention deficit hyperactivity disorder (ADHD). Eur Arch Paediatr Dent. 2018 Apr;19(2):91-97. doi: 10.1007/s40368-018-0330-3. Epub 2018 Mar 14. PMID 29542042
- [Background] Avsar A, Akbas S, Ataibis T. Traumatic dental injuries in children with attention deficit/hyperactivity disorder. Dent Traumatol. 2009 Oct;25(5):484-9. doi: 10.1111/j.1600-9657.2009.00792.x. Epub 2009 Jun 1. PMID 19496799
- [Background] Blomqvist M, Holmberg K, Fernell E, Dahllof G. A retrospective study of dental behavior management problems in children with attention and learning problems. Eur J Oral Sci. 2004 Oct;112(5):406-11. doi: 10.1111/j.1600-0722.2004.00150.x. PMID 15458498
- [Background] Sujlana A, Dang R. Dental care for children with attention deficit hyperactivity disorder. J Dent Child (Chic). 2013 May-Aug;80(2):67-70. PMID 24011294
- [Background] Marsh PD. Dental plaque: biological significance of a biofilm and community life-style. J Clin Periodontol. 2005;32 Suppl 6:7-15. doi: 10.1111/j.1600-051X.2005.00790.x. PMID 16128825
- [Background] Nishihara T, Koseki T. Microbial etiology of periodontitis. Periodontol 2000. 2004;36:14-26. doi: 10.1111/j.1600-0757.2004.03671.x. No abstract available. PMID 15330940
- [Background] Schmidt JC, Zaugg C, Weiger R, Walter C. Brushing without brushing?--a review of the efficacy of powered toothbrushes in noncontact biofilm removal. Clin Oral Investig. 2013 Apr;17(3):687-709. doi: 10.1007/s00784-012-0836-8. Epub 2012 Sep 23. PMID 23001187
- [Background] Turgut MD, Keceli TI, Tezel B, Cehreli ZC, Dolgun A, Tekcicek M. Number, length and end-rounding quality of bristles in manual child and adult toothbrushes. Int J Paediatr Dent. 2011 May;21(3):232-9. doi: 10.1111/j.1365-263X.2010.01102.x. Epub 2010 Oct 21. PMID 20961341
- [Background] Slot DE, Wiggelinkhuizen L, Rosema NA, Van der Weijden GA. The efficacy of manual toothbrushes following a brushing exercise: a systematic review. Int J Dent Hyg. 2012 Aug;10(3):187-97. doi: 10.1111/j.1601-5037.2012.00557.x. Epub 2012 Jun 6. PMID 22672101
- [Background] Thomassen TMJA, Van der Weijden FGA, Slot DE. The efficacy of powered toothbrushes: A systematic review and network meta-analysis. Int J Dent Hyg. 2022 Feb;20(1):3-17. doi: 10.1111/idh.12563. Epub 2021 Dec 31. PMID 34877772
- [Background] Rosema N, Slot DE, van Palenstein Helderman WH, Wiggelinkhuizen L, Van der Weijden GA. The efficacy of powered toothbrushes following a brushing exercise: a systematic review. Int J Dent Hyg. 2016 Feb;14(1):29-41. doi: 10.1111/idh.12115. Epub 2014 Dec 25. PMID 25545231
- [Background] Elkerbout TA, Slot DE, Rosema NAM, Van der Weijden GA. How effective is a powered toothbrush as compared to a manual toothbrush? A systematic review and meta-analysis of single brushing exercises. Int J Dent Hyg. 2020 Feb;18(1):17-26. doi: 10.1111/idh.12401. Epub 2019 Jul 23. PMID 31050195
- [Background] Davidovich E, Shafir S, Shay B, Zini A. Plaque Removal by a Powered Toothbrush Versus a Manual Toothbrush in Children: A Systematic Review and Meta-Analysis. Pediatr Dent. 2020 Jul 15;42(4):280-287. PMID 32847667
- [Background] Zimmer S, Didner B, Roulet JF. Clinical study on the plaque-removing ability of a new triple-headed toothbrush. J Clin Periodontol. 1999 May;26(5):281-5. doi: 10.1034/j.1600-051x.1999.260503.x. PMID 10355617
- [Background] Garcia-Godoy F, Marcushamer M, Cugini M, Warren PR. The safety and efficacy of a children's power toothbrush and a manual toothbrush in 6-11 year-olds. Am J Dent. 2001 Aug;14(4):195-9. PMID 11699736
- [Background] Silverman J, Rosivack RG, Matheson PB, Houpt MI. Comparison of powered and manual toothbrushes for plaque removal by 4- to 5-year-old children. Pediatr Dent. 2004 May-Jun;26(3):225-30. PMID 15185803
- [Background] Erbe C, Klees V, Braunbeck F, Ferrari-Peron P, Ccahuana-Vasquez RA, Timm H, Grender J, Cunningham P, Adam R, Wehrbein H. Comparative assessment of plaque removal and motivation between a manual toothbrush and an interactive power toothbrush in adolescents with fixed orthodontic appliances: A single-center, examiner-blind randomized controlled trial. Am J Orthod Dentofacial Orthop. 2019 Apr;155(4):462-472. doi: 10.1016/j.ajodo.2018.12.013. PMID 30935601
- [Background] Sandstrom A, Cressey J, Stecksen-Blicks C. Tooth-brushing behaviour in 6-12 year olds. Int J Paediatr Dent. 2011 Jan;21(1):43-9. doi: 10.1111/j.1365-263X.2010.01080.x. PMID 20659179
- [Background] Yaacob M, Worthington HV, Deacon SA, Deery C, Walmsley AD, Robinson PG, Glenny AM. Powered versus manual toothbrushing for oral health. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD002281. doi: 10.1002/14651858.CD002281.pub3. PMID 24934383
- [Background] Dogan MC, Alacam A, Asici N, Odabas M, Seydaoglu G. Clinical evaluation of the plaque-removing ability of three different toothbrushes in a mentally disabled group. Acta Odontol Scand. 2004 Dec;62(6):350-4. doi: 10.1080/00016350410010054. PMID 15848980
- [Background] Droubi L, Laflouf M, Alkurdi S, Sauro S, Mancino D, Haikel Y, Kharouf N. Does Customized Handle Toothbrush Influence Dental Plaque Removal in Children with Down Syndrome? A Randomized Controlled Trial. Healthcare (Basel). 2021 Aug 30;9(9):1130. doi: 10.3390/healthcare9091130. PMID 34574905
- [Background] Davidovich E, Ccahuana-Vasquez RA, Timm H, Grender J, Cunningham P, Zini A. Randomised clinical study of plaque removal efficacy of a power toothbrush in a paediatric population. Int J Paediatr Dent. 2017 Nov;27(6):558-567. doi: 10.1111/ipd.12298. Epub 2017 May 11. PMID 28494116
- [Background] Grossman E, Proskin H. A comparison of the efficacy and safety of an electric and a manual children's toothbrush. J Am Dent Assoc. 1997 Apr;128(4):469-74. doi: 10.14219/jada.archive.1997.0232. PMID 9103798
- [Background] Davidovich E, Ccahuana-Vasquez RA, Timm H, Grender J, Zini A. Randomised clinical study of plaque removal efficacy of an electric toothbrush in primary and mixed dentition. Int J Paediatr Dent. 2021 Sep;31(5):657-663. doi: 10.1111/ipd.12753. Epub 2021 Feb 14. PMID 33225464
- [Background] Mafla AC, Benavides RJ, Meyer P, Giraudeau N, Schwendicke F. Association of children's toothbrushing and fine motor skills: a cross-sectional study. Braz Oral Res. 2022 Jul 11;36:e103. doi: 10.1590/1807-3107bor-2022.vol36.0103. eCollection 2022. PMID 35830146
- [Background] Hidas A, Birman N, Noy AF, Shapira J, Matot I, Steinberg D, Moskovitz M. Salivary bacteria and oral health status in medicated and non-medicated children and adolescents with attention deficit hyperactivity disorder (ADHD). Clin Oral Investig. 2013 Nov;17(8):1863-7. doi: 10.1007/s00784-012-0876-0. Epub 2012 Nov 8. PMID 23135427
- [Background] Pitcher TM, Piek JP, Hay DA. Fine and gross motor ability in males with ADHD. Dev Med Child Neurol. 2003 Aug;45(8):525-35. doi: 10.1017/s0012162203000975. PMID 12882531
- [Background] Hidas A, Noy AF, Birman N, Shapira J, Matot I, Steinberg D, Moskovitz M. Oral health status, salivary flow rate and salivary quality in children, adolescents and young adults with ADHD. Arch Oral Biol. 2011 Oct;56(10):1137-41. doi: 10.1016/j.archoralbio.2011.03.018. Epub 2011 Apr 22. PMID 21514566
- [Background] Clinical practice guideline: diagnosis and evaluation of the child with attention-deficit/hyperactivity disorder. American Academy of Pediatrics. Pediatrics. 2000 May;105(5):1158-70. doi: 10.1542/peds.105.5.1158. PMID 10836893
- [Background] Vasileva M, Graf RK, Reinelt T, Petermann U, Petermann F. Research review: A meta-analysis of the international prevalence and comorbidity of mental disorders in children between 1 and 7 years. J Child Psychol Psychiatry. 2021 Apr;62(4):372-381. doi: 10.1111/jcpp.13261. Epub 2020 May 20. PMID 32433792
- [Background] Zorlu A, Unlu G, Cakaloz B, Zencir M, Buber A, Isildar Y. The Prevalence and Comorbidity Rates of ADHD Among School-Age Children in Turkey. J Atten Disord. 2020 Jul;24(9):1237-1245. doi: 10.1177/1087054715577991. Epub 2015 Apr 6. PMID 25846229
- [Background] Millichap JG. Etiologic classification of attention-deficit/hyperactivity disorder. Pediatrics. 2008 Feb;121(2):e358-65. doi: 10.1542/peds.2007-1332. PMID 18245408
- [Background] Palladino VS, McNeill R, Reif A, Kittel-Schneider S. Genetic risk factors and gene-environment interactions in adult and childhood attention-deficit/hyperactivity disorder. Psychiatr Genet. 2019 Jun;29(3):63-78. doi: 10.1097/YPG.0000000000000220. PMID 30741787
- [Background] Caye A, Swanson JM, Coghill D, Rohde LA. Treatment strategies for ADHD: an evidence-based guide to select optimal treatment. Mol Psychiatry. 2019 Mar;24(3):390-408. doi: 10.1038/s41380-018-0116-3. Epub 2018 Jun 28. PMID 29955166
- [Background] Sharma A, Couture J. A review of the pathophysiology, etiology, and treatment of attention-deficit hyperactivity disorder (ADHD). Ann Pharmacother. 2014 Feb;48(2):209-25. doi: 10.1177/1060028013510699. Epub 2013 Nov 1. PMID 24259638
- [Background] Sonuga-Barke EJ, Brandeis D, Cortese S, Daley D, Ferrin M, Holtmann M, Stevenson J, Danckaerts M, van der Oord S, Dopfner M, Dittmann RW, Simonoff E, Zuddas A, Banaschewski T, Buitelaar J, Coghill D, Hollis C, Konofal E, Lecendreux M, Wong IC, Sergeant J; European ADHD Guidelines Group. Nonpharmacological interventions for ADHD: systematic review and meta-analyses of randomized controlled trials of dietary and psychological treatments. Am J Psychiatry. 2013 Mar;170(3):275-89. doi: 10.1176/appi.ajp.2012.12070991. PMID 23360949
- [Background] Subcommittee on Attention-Deficit/Hyperactivity Disorder; Steering Committee on Quality Improvement and Management; Wolraich M, Brown L, Brown RT, DuPaul G, Earls M, Feldman HM, Ganiats TG, Kaplanek B, Meyer B, Perrin J, Pierce K, Reiff M, Stein MT, Visser S. ADHD: clinical practice guideline for the diagnosis, evaluation, and treatment of attention-deficit/hyperactivity disorder in children and adolescents. Pediatrics. 2011 Nov;128(5):1007-22. doi: 10.1542/peds.2011-2654. Epub 2011 Oct 16. PMID 22003063
- [Background] Chau YC, Lai KY, McGrath CP, Yiu CK. Oral health of children with attention deficit hyperactivity disorder. Eur J Oral Sci. 2017 Feb;125(1):49-54. doi: 10.1111/eos.12323. Epub 2016 Dec 30. PMID 28035689
- [Background] Blomqvist M, Ahadi S, Fernell E, Ek U, Dahllof G. Dental caries in adolescents with attention deficit hyperactivity disorder: a population-based follow-up study. Eur J Oral Sci. 2011 Oct;119(5):381-5. doi: 10.1111/j.1600-0722.2011.00844.x. Epub 2011 Aug 12. PMID 21896055
- [Background] Ehlers V, Callaway A, Wantzen S, Patyna M, Deschner J, Azrak B. Oral health of children and adolescents with or without attention deficit hyperactivity disorder (ADHD) living in residential care in rural Rhineland-Palatinate, Germany. BMC Oral Health. 2019 Nov 25;19(1):258. doi: 10.1186/s12903-019-0948-5. PMID 31766996
- [Background] Cortese S, Moreira Maia CR, Rohde LA, Morcillo-Penalver C, Faraone SV. Prevalence of obesity in attention-deficit/hyperactivity disorder: study protocol for a systematic review and meta-analysis. BMJ Open. 2014 Mar 18;4(3):e004541. doi: 10.1136/bmjopen-2013-004541. PMID 24643169
- [Background] Dursun OB, Sengul F, Esin IS, Demirci T, Yucel N, Omezli MM. Mind Conduct disorders in children with poor oral hygiene habits and attention deficit hyperactivity disorder in children with excessive tooth decay. Arch Med Sci. 2016 Dec 1;12(6):1279-1285. doi: 10.5114/aoms.2016.59723. Epub 2016 May 5. PMID 27904519
- [Background] Kohlboeck G, Heitmueller D, Neumann C, Tiesler C, Heinrich J, Heinrich-Weltzien R, Hickel R, Koletzko S, Herbarth O, Kuhnisch J; GINIplus Study Group, LISAplus Study Group. Is there a relationship between hyperactivity/inattention symptoms and poor oral health? Results from the GINIplus and LISAplus study. Clin Oral Investig. 2013 Jun;17(5):1329-38. doi: 10.1007/s00784-012-0829-7. Epub 2012 Aug 29. PMID 22927131